CLINICAL TRIAL: NCT05785104
Title: Effect of Muscle Energy Technique Versus Myofascial Release on Cervical and Lumbar Pain in Premenopausal Women With Fibromyalgia
Brief Title: Effect of Muscle Energy Technique Versus Myofascial Release on Cervical and Lumbar Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Samar Ahmed Abd EL Salam Negm, Samar Ahmed Abd El Salam Negm, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 012/004046
Record Dates: First submitted 2023-03-14; First posted 2023-03-27 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Lumbar Pain Syndrome; Cervical Pain
Keywords: Cervical pain,lumbar pain,fibromyalgia
MeSH Terms: conditions — Somatoform Disorders; Neck Pain | interventions — Myofascial Release Therapy

STUDY DESIGN:
Intervention Model Description: Two groups, one group will be treated by muscle energy technique and other will be treated by myofascial release
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofascial release (Experimental): The patients will receive myofascial release technique on cervical and lumbar regions three times per week for four weeks
  Interventions: Other: Myofascial release
- Muscle energy technique (Experimental): The patients will receive muscle energy technique for cervical and lumbar regions three times per week for four weeks
  Interventions: Other: Muscle energy technique

INTERVENTIONS:
Other: Myofascial release — Is Facilitation of mechanical and neurological adaptive capacity as integrated through the Myofascial system
  Arms: Myofascial release
Other: Muscle energy technique — Is manual therapy procedure that involves alternating periods of resisted muscle contraction and assisted stretching
  Arms: Muscle energy technique

SUMMARY:
The aim of the study is to determine the effect of muscle energy technique versus myofascial release on cervical and lumbar pain in premenopausal women with fibromyalgia

DETAILED DESCRIPTION:
Fibromyalgia is an idiopathic, non articular pain syndrome with generalized tender points. It is multisystem disease characterized by sleep disturbance and fatigue. It affect 5% of the world population. The incidence is higher in women than in men. And the age is between 30 and 35 years old.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women with fibromyalgia
* Ages ranges between 30 - 45 years old
* Body mass index < 35 kg/m2
* All are medically stable

Exclusion Criteria:

* specific cervical and lumbar pain
* Smokers
* Pregnant women
* Medically unstable
* Postmenopausal women

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia impact questionnaire | Four weeks
  Used to assess health related quality of life before and after the treatment, maximum score means worse outcome
Visual analogue scale | Four weeks
  Used to assess the severity of cervical and lumbar pain of each premenopausal women in both groups before and after the treatment, maximum score means worse outcome
Active range of motion of cervical and lumbar regions | Four weeks
  Measurement of active flexion, extension, lateral flexion in cervical and lumbar regions before and after the treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes